CLINICAL TRIAL: NCT06803537
Title: Three-Year Clinical Performance of Fiber-reinforced Versus Indirect Resin Composite Posterior Restorations
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A02071221
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-01

CONDITIONS: Occlusal Caries; Proximal Caries
Keywords: fiber-reinforced composite; indirect lab composite; posterior restorations

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fiber-reinforced composite (Active Comparator)
  Interventions: Other: indirect lab composite; Other: Conventional resin composite
- Indirect lab composite (Active Comparator)
  Interventions: Other: Fiber-reinforced composite; Other: Conventional resin composite
- Conventional microhybrid resin composite (Active Comparator)
  Interventions: Other: Fiber-reinforced composite; Other: indirect lab composite

INTERVENTIONS:
Other: Fiber-reinforced composite — short fiber-reinforced composite used as base covered by conventional composite
  Arms: Conventional microhybrid resin composite; Indirect lab composite
Other: indirect lab composite — indirect lab processed resin composite inlay restorations
  Arms: Conventional microhybrid resin composite; Fiber-reinforced composite
Other: Conventional resin composite — conventional microhybrid resin composite posterior restorations
  Arms: Fiber-reinforced composite; Indirect lab composite

SUMMARY:
This study aimed to perform a comparison between the clinical performance of short fiber-reinforced composite and indirect lab composite restorations in posterior dentition.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 20-35 year from both genders.
2. Good oral hygiene: patients with low and moderate caries risk (according to Caries management by caries risk assessment CAMBRA sheets) were enrolled in this study.
3. The visual examination should reveal the presence of a minimum of three primary occlusal or proximal caries (Black Class I and II) with a severity score of 4 or 5 according to the International Caries Detection and Assessment System (ICDAS).
4. The carious teeth must exhibit vitality and do not display periapical radiolucency as evaluated by periapical radiography.
5. The selected teeth must be under stable occlusion.

Exclusion Criteria:

1. Uncontrolled systemic disease
2. Extremely poor oral hygiene
3. Chronic periodontitis
4. Heavy bruxism
5. Cavities with a buccolingual width exceeding two-thirds of the intercuspal distance or requiring cusp covering.
6. Patients undergoing orthodontic procedures.
7. Patients unable to attend the scheduled recall appointments.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
FDI criteria for evaluation | Three years follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura university, Al Mansurah, Dakahlia Governorate, Egypt